CLINICAL TRIAL: NCT02190175
Title: Multicentre Non Interventional Study in the Management of Atrial Fibrillation With Flecainide
Brief Title: Management of Atrial Fibrillation With Flecainide : the AFFLEC Study
Status: Completed | Type: Observational
Sponsor: Hellenic Cardiovascular Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: AFFLEC
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicentre non interventional observational study with the objective to follow up patients with atrial fibrillation who based on current indications are treated with per os flecainide , for cardiac pulse maintenance.

DETAILED DESCRIPTION:
the study objectives are

* record safety and efficiency of flecainide as antiarrythmic treatment in atrial fibrillation
* study of flecainide in ST interval

ELIGIBILITY:
Inclusion Criteria:

* patients with history of atrial fibrillation
* patients able to give informed consent

Exclusion Criteria:

* patients with coronary disease or other cardiopathy with left heart champer affected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of atrial fibrillation who are under treatment with per os flecainide
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ST interval and repolarization measures of myocardia in patients under treatment of flecainide | 6months

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Erythros Stavros Hospital, Athens
  - University Hospital of Larisa, Larissa
  - AHEPA University Hospital, Thessaloniki